CLINICAL TRIAL: NCT05794620
Title: Faecal Microbiota Analysis in Neurotypical and Autism Syndrome Disorder Siblings: FAMILY
Brief Title: Faecal Microbiota Analysis in Neurotypical and Autism Syndrome Disorder Siblings
Acronym: FAMILY
Status: Completed | Type: Observational
Sponsor: East Suffolk and North Essex NHS Foundation Trust (Other)
Collaborators: Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Other Study IDs: 22/045
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Faecal samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Autism: A child with a diagnosis of Autism
  Interventions: Other: Stool sample
- Neurotypical siblings: A full sibling of the child with Autism
  Interventions: Other: Stool sample

INTERVENTIONS:
Other: Stool sample — Stool sample

SUMMARY:
This study aims to accurately characterise the gut microbiota composition of faeces of children with ASD and compare it with the gut microbiota composition of their neurotypical siblings. In addition it aims to also characterise the metagenome and metabolome of the faeces of both ASD and neurotypical siblings.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes who are diagnosed with ASD and under the care of ESNEFT who have a neurotypical sibling (either full or half sibling), who share their living environment. This is due to the study requiring stool samples that are from siblings, to control for genes and environment where possible.
* Aged 3 years to 10 years old (at time of consent)
* Parent/guardian able to consent to participate
* Parent/guardian able to complete required surveys (or with accommodated adjustments)

Exclusion Criteria:

* Use of antibiotics in the previous 4 weeks
* Not under the care of ESNEFT
* Children <3 years old and >10 years old
* Children that don't have half or full siblings
* Parent/guardian unable to provide informed consent or complete surveys, despite reasonable adjustments being implemented

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with ASD
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Gut microbiota | 0 weeks
  Gut microbiota composition of faeces of children with ASD

OTHER OUTCOMES:
Gut microbiota | 6 weeks
  Gut microbiota composition of faeces of children with ASD

CONTACTS AND LOCATIONS:
Overall Officials: Ben Marlow, Principal Investigator — East Suffolk and North Essex NHS Foundation Trust
Locations (1):
- East Suffolk and North Essex Nhs Foundation Trust, Colchester, United Kingdom